CLINICAL TRIAL: NCT02491944
Title: A Phase I, Open-label, Single Dose, Single-Centre Study to Assess the Absolute Bioavailability of a Single Oral Dose of AZD9291 With Respect to an Intravenous Microdose of [14C]AZD9291 in Healthy Male Subjects
Brief Title: A Phase I, Open-label Study to Assess Bioavailability of a Single Oral Dose of AZD9291 vs an IV Dose of [14C]AZD9291
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00020
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioavailability of AZD9291 (Experimental): To assess the absolute bioavailability of a single oral dose of AZD9291 with respect to an intravenous microdose of [14C]AZD9291
  Interventions: Drug: AZD9291; Drug: [14C]AZD9291

INTERVENTIONS:
Drug: AZD9291 — Single oral dose of 80 mg AZD9291 tablet on Day 1 administered orally with 240 mL water following an overnight fast.
Drug: [14C]AZD9291 — Each healthy male subject will also receive a single, radiolabeled, 100 μg dose of [14C] AZD9291 administered as an IV microdose infusion starting at 5 hours and 45 minutes after receiving the oral dose.

SUMMARY:
The Sponsor is developing the study drug, AZD9291, for the potential treatment of nonsmall cell lung cancer. Lung cancer has been the most common cancer in the world for several decades and represents 12.8% of all new cancer cases in 2008.

The purpose of this study is to see how much AZD9291 is taken up by the body when dosed by mouth (tablet) compared to when the study drug is dosed once by injection directly into the vein (intravenously). The dose given directly into the vein will be radiolabelled. This means that the test drug has a radioactive component which helps us to track where the drug is in the body. This allows us to detect the differences between the tablet and the intravenous dose.

The study will be performed in 12 healthy male subjects aged 18-65 years. On Day 1, subjects will be dosed with a single oral dose of 80 milligrams AZD9291 tablet followed by 100 micrograms [14C] AZD9291 dosed as an intravenous microdose beginning 5 hours and 45 minutes after the oral dose has been administered. Subjects will remain in the study centre until after the 120 hour post-dose blood sample is obtained and will return to the clinic for further visits on Day 8, 10, 15 and 22 for pharmacokinetic and safety assessments.

DETAILED DESCRIPTION:
The study is a Phase I, open label, single dose, single centre study performed in 12 healthy male subjects aged 18 to 65 years, inclusive. This study will assess the absolute bioavailability of AZD9291 and evaluate the PK parameters following a single oral dose of AZD9291 and a radiolabelled IV microdose of AZD9291 in healthy male subjects. Oral AZD9291and [14C] AZD9291 intravenous solution are referred to as the investigational products in this study.

A screening visit (Visit 1) to assess the eligibility of the healthy male subjects will occur within 28 days of the administration of the investigational product. Screening assessments will include evaluation of opthalmological assessments, clinical chemistry, haematology, urinalysis, a physical examination, vital signs, 12-lead electrocardiograms (ECGs), medical and surgical history, screening for drugs of abuse, alcohol, hepatitis B and C, and HIV, and recording of concomitant medications and Adverse Events. Study related procedures will only be performed after signing of the Informed Consent Form.

The healthy male subjects will be admitted to the study centre the day before administration of the investigational product (Day 1; Visit 2). On Day 1 (Visit 2), subjects will be dosed with a single oral dose of 80 mg AZD9291 tablet followed by 100 μg [14C] AZD9291 dosed as an IV microdose beginning 5 hours and 45 minutes after the oral dose has been administered. The IV microdose will be infused over 15 minutes and the end of the infusion will be co incidental with median oral tmax (ie, estimated tmax is 6 hours).

The subjects will remain in the study centre until the 120 hour post dose PK blood sample is obtained. Ambulatory visits will occur on Days 8 (Visit 3), 10 (Visit 4), 15 (Visit 5) and 22 (Visit 6) for PK and safety assessments. A follow up visit (Visit 7) will occur 21 to 28 days after discharge (Days 27 - 34) from the study centre and will include routine safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed dated, written informed consent.
2. Healthy male aged 18 to 65 yrs with suitable veins for blood sampling
3. BMI: 19 and 32 kg/m2 inclusive, weight at least 50 kg and no more than 100 kg, inclusive.
4. At screening, calculated creatinine clearance ≥50 mL/min using Cockcroft Gault formula.
5. Willing to use defined methods of contraception
6. Willing and able to comply with study procedures, restrictions and requirements.
7. Provision of informed consent for genetic research. Declining genetic research will not exclude subjects from other aspects of study.

Exclusion Criteria:

1. Involvement in planning and/or conduct of study.
2. Subjects previously enrolled in this study.
3. History of clinically significant disease or disorder which, either puts subject at risk because of participation in study, or influences results or subject's ability to participate in study.
4. History or presence of condition known to interfere with ADME of drugs.
5. Any clinically significant abnormalities in physical examination, as judged by PI.
6. Acute illness, surgical procedures, or trauma from within 2 wks before screening until first admin of investigational product (IMP).
7. Subjects who have received live or live-attenuated vaccine in 2 wks prior to IMP admin.
8. Subjects with active malignancy or neoplastic disease in previous 12 mths.
9. A suspected/manifested infection according to IATA Categories A and B.
10. Positive screening tests for serum hepatitis B surface antigen, hepatitis C antibody, or HIV.
11. Any clinically important abnormalities in rhythm, conduction, or morphology of resting 12-lead ECG, QT interval >470 ms.
12. Known or suspected history of significant drug abuse.
13. Positive screen for drugs of abuse or cotinine at screening or positive screen for alcohol, drugs of abuse, or cotinine on admission to centre prior to first admin of IMP.
14. History of alcohol abuse or excessive intake of alcohol, defined as regular weekly intake of more than 21 units of alcohol in men
15. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by PI, or history of hypersensitivity to AZD9291, its excipients, or drugs with a similar chemical structure or class.
16. Use of any prescribed or non-prescribed medication, including drugs during the 4 wks (or longer depending on the medication's half-life) prior to admin of AZD9291 is not permitted. Occasional use of paracetamol and adrenergic nasal spray for relief of nasal congestion is permitted at the discretion of the PI. Exceptions as agreed by PI and sponsor's medical monitor if do not interfere with aims of study.
17. Use of drugs with enzyme inducing properties such as St John's Wort within 4 wks prior to IMP administration.
18. Any intake of grapefruit, grapefruit juice, Seville oranges or products containing these fruit within 7 days of first admin of IMP.
19. Blood donation within 1 mth of screening or any blood donation/blood loss greater than 500 mL during 3 mths prior to screening.
20. Subjects who received another NCE or participated in any other clinical study (including methodology studies where no drugs were given) within 3 mths of first admin of IMP
21. Judgment by PI that subject should not participate in study if subject is considered unlikely to comply with study procedures, restrictions, and requirements.
22. Ongoing or planned inpatient surgery, dental procedure, or hospitalisation during study
23. Radiation exposure exceeding 5 mSv in last 12 mths or 10 mSv in last 5 yrs.
24. Admin of any amount of a [14C]-labelled compound within last 12 mths.
25. Used of nicotine products (including cigarettes) within previous 3 mths.
26. Judgment by PI that subject would not be able to understand or cooperate with requirements of study.
27. Previous bone marrow transplant
28. Blood transfusion within 120 days of genetic sample collection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Collier, MBChB, FFPM, Dip Stats (OU), Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Research Site, Nottingham, United Kingdom

REFERENCES:
- [Derived] Vishwanathan K, So K, Thomas K, Bramley A, English S, Collier J. Absolute Bioavailability of Osimertinib in Healthy Adults. Clin Pharmacol Drug Dev. 2019 Feb;8(2):198-207. doi: 10.1002/cpdd.467. Epub 2018 Apr 23. PMID 29683562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 10 July 2015; Last subject last visit: 26 August 2015. This study was conducted in a single study centre in the UK.
Pre-assignment Details: 27 subjects were enrolled (signed informed consent). Subjects were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 17 subjects were enrolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment. The remaining 10 subjects received treatment.
Groups:
- AZD9291 and [14C]AZD9291: Single oral dose of 80 mg AZD9291 tablet on Day 1 and a single, radiolabeled, 100 μg dose of [14C] AZD9291 administered as an IV microdose infusion starting at 5 hours and 45 minutes after receiving the oral dose.
Period: Overall Study
Arm/Group | AZD9291 and [14C]AZD9291
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Oral Bioavailability
Description: Absolute bioavailability of AZD9291 will be calculated from area under the plasma concentration versus time curve (AUC) of the oral dose of AZD9291 / AUC of the IV dose of [14C]AZD9291 x IV dose/Oral dose x 100
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 5:45, 5:52, 6, 6:05, 6:10, 6:20, 6:25, 6:30, 7, 8, 9, 10, 12, 14, 16, 18, 24, 30, 48, 72, 120, 168, 216, 336 and 504 hours relative to the oral dose.
Population: PK analysis set included all healthy male subjects who received at least 1 dose of AZD9291 and have at least 1 post-dose PK measurement without important protocol deviations/violations or events thought to significantly affect the PK of AZD9291.
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
Percentage | 69.75 [66.71 to 72.92]

2. Secondary Outcome: AUC for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: Pharmacokinetic (PK) profile of the oral dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from zero to infinity for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*h
  AZD9291 | 6791 (27.6)
  AZ5104 | 694.5 (37.6)
  AZ7550 | 602.5 (28.6)

3. Secondary Outcome: AUC(0-24) for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: Pharmacokinetic (PK) profile of the oral dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to 24 hours (AUC 0-24) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*h
  AZD9291 | 1963 (26.6)
  AZ5104 | 113.7 (40.1)
  AZ7550 | 75.38 (33.8)

4. Secondary Outcome: AUC(0-120) for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: Pharmacokinetic (PK) profile of the oral dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to 120 hours (AUC 0-120) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*h
  AZD9291 | 5545 (25.3)
  AZ5104 | 512.9 (37.2)
  AZ7550 | 361.8 (28.8)

5. Secondary Outcome: AUC(0-t) for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: Pharmacokinetic (PK) profile of the oral dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to the last quantifiable concentration (AUC 0-t) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*h
  AZD9291 | 6770 (27.6)
  AZ5104 | 684.4 (37.6)
  AZ7550 | 591.2 (29.0)

6. Secondary Outcome: Cmax for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: PK profile of the oral dose of AZD9291 in terms of the maximum observed plasma concentration (Cmax) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM
  AZD9291 | 118.0 (28.1)
  AZ5104 | 6.187 (38.0)
  AZ7550 | 4.302 (34.3)

7. Secondary Outcome: Tmax for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: PK profile of the oral dose of AZD9291 in terms of the time to maximum observed plasma concentration (Tmax) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
hours
  AZD9291 | 7.01 (28.1) [6.00 to 10.00]
  AZ5104 | 12.00 (38.0) [6.00 to 48.07]
  AZ7550 | 11.03 (34.3) [8.00 to 48.00]

8. Secondary Outcome: t1/2,λz for AZD9291 and it's Metabolites AZ5104 and AZ7550
Description: PK profile of the oral dose of AZD9291 in terms of the elimination half life (t1/2,λz) for AZD9291 and it's metabolites AZ5104 and AZ7550.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
hours
  AZD9291 | 59.72 (4.257) [6.00 to 10.00]
  AZ5104 | 52.59 (7.355) [6.00 to 48.07]
  AZ7550 | 72.58 (11.86) [8.00 to 48.00]

9. Secondary Outcome: CL/F for AZD9291
Description: PK profile of the oral dose of AZD9291 in terms of apparent total body clearance of drug from plasma after extravascular administration(CL/F) for AZD9291.
Time Frame: Samples taken at pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 504 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
L/h | 24.40 (6.979) [6.00 to 10.00]

10. Secondary Outcome: AUC for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from zero to infinity for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: Samples taken pre-dose, during the infusion, immediately at the end of infusion and then at 5, 10, 20, 25 and 30 minutes and 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 42, 66, 114, 162, 210, 330 and 498 hours after the end of the infusion.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*eq*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*eq*h
  [14C]AZD9291 | 12.12 (22.8)
  [14C]AZ5104 | 1.247 (26.8)
  [14C]AZ7550 | 1.177 (19.9)

11. Secondary Outcome: AUC(0-24) for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to 24 hours (AUC 0-24) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*eq*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*eq*h
  [14C]AZD9291 | 3.463 (21.6)
  [14C]AZ5104 | 0.1172 (36.1)
  [14C]AZ7550 | 0.08919 (28.5)

12. Secondary Outcome: AUC(0-120) for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to 120 hours (AUC 0-120) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*eq*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*eq*h
  [14C]AZD9291 | 9.551 (22.1)
  [14C]AZ5104 | 0.7450 (34.4)
  [14C]AZ7550 | 0.5292 (28.9)

13. Secondary Outcome: AUC(0-t) for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of Area under the plasma concentration - time curve (AUC) from time zero to the last quantifiable concentration (AUC 0-t) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*eq*h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*eq*h
  [14C]AZD9291 | 11.64 (25.7)
  [14C]AZ5104 | 0.8802 (44.2)
  [14C]AZ7550 | 0.6899 (38.1)

14. Secondary Outcome: Cmax for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of the maximum observed plasma concentration (Cmax) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*eq
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
nM*eq
  [14C]AZD9291 | 0.5762 (68.6)
  [14C]AZ5104 | 0.008309 (36.1)
  [14C]AZ7550 | 0.005751 (34.2)

15. Secondary Outcome: Tmax for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of the the time to maximum observed plasma concentration (Tmax) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
hours
  [14C]AZD9291 | 0.25 (68.6) [0.12 to 0.67]
  [14C]AZ5104 | 42.25 (36.1) [12.25 to 66.37]
  [14C]AZ7550 | 33.27 (34.2) [18.27 to 66.37]

16. Secondary Outcome: t1/2,λz for [14C]AZD9291 and it's Metabolites [14C]AZ5104 and [14C]AZ7550
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of the elimination half life (t1/2,λz) for [14C]AZD9291 and it's metabolites [14C]AZ5104 and [14C]AZ7550.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
hours
  [14C]AZD9291 | 54.93 (9.032) [0.12 to 0.67]
  [14C]AZ5104 | 68.35 (15.73) [12.25 to 66.37]
  [14C]AZ7550 | 99.69 (29.33) [18.27 to 66.37]

17. Secondary Outcome: CL for [14C]AZD9291
Description: Pharmacokinetic (PK) profile of the IV dose of AZD9291 in terms of total body clearance of drug from plasma after intravascular administration (CL) for [14C]AZD9291.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AZD9291 and [14C]AZD9291
Number analyzed (Participants) | 10
L/h | 16.84 (3.941) [0.12 to 0.67]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 30 days starting from the dosing day
Description: Regular investigator assessment at study visits.
Arm/Group | AZD9291 and [14C]AZD9291
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 and [14C]AZD9291 (N=10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.